CLINICAL TRIAL: NCT05659186
Title: A Phase II Study of the Efficacy and Safety of PD-1 Inhibitor and Anlotinib Combined With Multimodal Radiotherapy in the Second-line Treatment of Recurrent or Metastatic Anaplastic Thyroid Cancer
Brief Title: PD-1 Inhibitor and Anlotinib Combined With Multimodal Radiotherapy in Recurrent or Metastatic Anaplastic Thyroid Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR2100054455
Record Dates: First submitted 2022-12-08; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer; Immunotherapy; Radiotherapy; Anlotinib
MeSH Terms: conditions — Thyroid Neoplasms | interventions — tislelizumab; anlotinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental): Tislelizumab administration on day 1, and Anlotinib continuous administration from days 1 to 14， every three weeks Radiotherapy
  Interventions: Drug: Tislelizumab; Drug: Anlotinib; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Tislelizumab — 200mg IV Q3W
  Other Names: BGB-A317
Drug: Anlotinib — 12mg PO QD
  Other Names: AL3818
Radiation: Radiotherapy — Multimodal Radiotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PD-1 inhibitor and anlotinib combined with multimodal radiotherapy for the second-line treatment of recurrent or metastatic anaplastic thyroid cancer.

DETAILED DESCRIPTION:
Thyroid cancer (TC) is the most common malignant tumor of the endocrine system. It is more common in women and accounts for approximately 4% of all new malignancies in women. TC can be classified according to its pathological type: papillary carcinoma, follicular carcinoma, Hurthle cell carcinoma, medullary carcinoma, and anaplastic thyroid carcinoma (ATC). ATC is more aggressive than other types and tends to metastasize at an early stage. Although ATC accounts for only 1.6%-4% of all TC, the mortality rate is 14%-40%. According to the American Joint Committee on Cancer (AJCC) staging criteria, all ATC is considered stage IV once diagnosed, regardless of the size of the primary site or lymph node metastasis. Until now, the best treatment options for ATC have been unclear, and currently, a combination of treatment options is used. However, the efficiency of treatment is less than 15% and most patients experience recurrence and distant metastases. There is an urgent need for safe and effective treatment options for patients with ATC.

Radiotherapy, as one of the important local treatments, can reduce the tumor load and alleviate local symptoms. Several studies have demonstrated that radiotherapy can improve the prognosis of patients with ATC. The results of a meta-analysis covering 17 studies with a total of 1147 patients showed that postoperative radiotherapy improved the prognosis of patients with ATC compared to those who underwent surgery only. Meanwhile, the results of another large retrospective study showed that radiotherapy resulted in sustained local progression-free survival and overall survival in the treatment of patients with locally advanced ATC and that a radiotherapy dose of ≥60 Gy was an independent prognostic factor (p=0.01). The prognostic role of radiotherapy and different radiotherapy doses was also confirmed in another meta-analysis from the National Cancer Database (NCDB), which showed that patients with inoperable ATC may benefit from radiotherapy at higher irradiation doses (60-70 Gy vs 45-59.9 Gy). It can thus be seen that both operable and inoperable ATC patients, may benefit from radiotherapy and that the dose of radiotherapy may correlate with their survival benefit.

For the systemic treatment of patients with ATC, the NCCN guidelines recommend first-line regimens including paclitaxel combined with carboplatin, doxorubicin combined with doxorubicin, single-agent paclitaxel and single-agent doxorubicin, but patients with ATC respond poorly to treatment and there is no recommended optimal regimen for patients who develop recurrence or metastasis after first-line therapy. In recent years, PD-1/PD-L1 has been used in melanoma and a variety of other solid tumors have demonstrated promising efficacy. The results of a retrospective study in 2017 showed positive PD-1 expression in all specimens of the 16 ATC patients observed, while almost all patients (13/16) were positive for PD-L1 expression. In vitro experiments have also shown that PD-1 blockers can reinvigorate the cytotoxic effects of NK cells, thereby enhancing the killing effect on tumor cells. This lays the theoretical foundation for the use of PD-1/PD-L1 blockers in the treatment of ATC. Multi-target tyrosine kinase inhibitors have shown significant anti-tumor effects in a variety of tumor types, including thyroid cancer, by inhibiting angiogenic and proliferative signaling. Anrotinib is a small molecule multi-target complex kinase inhibitor developed in China and has been reported to be safe and effective in the treatment of patients with advanced refractory solid tumors. In addition to this, the anti-tumor activity of anrotinib in ATC has been In vivo and in vitro assays have demonstrated that anlotinib inhibits ATC cell proliferation and inhibits the migration of thyroid cancer cells in vitro and the growth of xenograft thyroid tumors in mice.

The findings suggest that there may be synergy between PD-1/PD-L1 blockers and complex kinase inhibitors and that PD-1/PD-L1 blockers may improve the tumor microenvironment in ATC, thereby increasing the efficacy of complex kinase inhibitors. This suggests that the combination of PD-1/PD-L1 blockers and complex kinase inhibitors may be an effective treatment option for ATC and that PD-1/PD-L1 blockers may improve resistance to complex kinase inhibitor therapy. PD-L1 blockers may improve the resistance that occurs with complex kinase inhibitor therapy. Meanwhile, the combination of PD-1/PD-L1 blockers with radiotherapy has been shown to have a synergistic effect in several studies. Radiotherapy combined with immunotherapy can activate specific T-cell immune responses and alter the suppressive effect of the tumor microenvironment on the immune system, resulting in durable anti-tumor activity. Combining radiotherapy with PD-1/PD-L1 blockers for the treatment of undifferentiated thyroid cancer may demonstrate better therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above.
2. Patients with pathologically confirmed Undifferentiated thyroid carcinoma and meet the following conditions:

   1. Were diagnosed with distant metastasis;
   2. Were intolerant to or failed first-line treatment.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
4. Expected life is greater than or equal to 12 weeks.
5. There is at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
6. Adequate organ and bone marrow function:

   1. Absolute neutrophil count ≥ 1.5 × 10^9/L, hemoglobin ≥ 80 g/L, platelets ≥ 80 × 10^9/L;
   2. ALT, AST and ALP < 2.5× upper limit of normal (ULN), total bilirubin ≤ 2×ULN; albumin≥ 2.8 g/dL；
   3. Creatinine clearance ≥ 60 ml/min;
   4. INR≤ 1.5, APTT≤ 1.5×ULN.
7. Written informed consent.

Exclusion Criteria:

1. Existing tumor-related hemorrhage。
2. History of other malignancies (except for the history of malignant tumors that have been cured and have not recurred within 5 years, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, in situ cervical cancer, and gastrointestinal mucosal cancer, etc.）
3. Have an active autoimmune disease requiring systemic treatment or a documented history of clinically severe autoimmune disease.
4. Any history of allergic disease, severe hypersensitivity reaction to drugs, or allergy to the study drug components.
5. Any prior therapy with:

   1. Toxicity from prior antitumor therapy has not recovered to ≤ CTCAE Version 5.0 Grade 1 or the level specified by the inclusion/exclusion criteria.
   2. Antitumor vaccine;
   3. Any active vaccine against infectious disease within 4 weeks prior to the first dose or planned during the study period;
   4. Major surgery or serious trauma within 4 weeks before the first dose;
6. With serious medical diseases, such as grade II and above cardiac dysfunction (NYHA criteria), ischemic heart disease, supraventricular or ventricular arrhythmia, poorly controlled diabetes mellitus, poorly controlled hypertension, echocardiographic ejection fraction < 50%, etc.
7. With interstitial pneumonitis, non-infectious pneumonitis, active pulmonary tuberculosis, or a history of pulmonary tuberculosis infection that was not controlled by treatment.
8. With hyperthyroidism, or organic thyroid disease.
9. With active infection, or unexplained fever during the screening period or 48 hours before the first dose.
10. With active hepatitis B or C, or known history of positive HIV test, or acquired immunodeficiency syndrome.
11. History of a clear neurological or psychiatric disorder.
12. History of drug abuse or alcohol abuse.
13. Women who are pregnant or breastfeeding, or have a reproductive plan from the screening period to 3 months after the end of the study, or have sex without contraceptive measures, or are unwilling to take appropriate contraceptive measures.
14. Received any investigational drug within 4 weeks prior to the first dose, or concurrently enrolled in another clinical trial.
15. Any other factors that are not suitable for inclusion in this study judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 60 months
  ORR is defined as the percentage of patients who achieve a response, which can either be complete response (complete disappearance of lesions) or partial response (reduction in the sum of maximal tumor diameters by at least 30% or more)

SECONDARY OUTCOMES:
Progress-Free Survival | Up to 60 months
  PFS is defined as the time from the administration of the first dose to first disease progression or death.
Overall Survival | Up to 60 months
  OS is defined as the time from the administration of the first dose to death.
Adverse events | Up to 60 months
  defined as the number of participants with adverse events using CTCAE Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Professor, Principal Investigator — West China Hospital
Locations (1):
- Xingchen Peng, Chengdu, Sichuan, China

REFERENCES:
- [Background] Lin B, Ma H, Ma M, Zhang Z, Sun Z, Hsieh IY, Okenwa O, Guan H, Li J, Lv W. The incidence and survival analysis for anaplastic thyroid cancer: a SEER database analysis. Am J Transl Res. 2019 Sep 15;11(9):5888-5896. eCollection 2019. PMID 31632557
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Haddad RI, Nasr C, Bischoff L, Busaidy NL, Byrd D, Callender G, Dickson P, Duh QY, Ehya H, Goldner W, Haymart M, Hoh C, Hunt JP, Iagaru A, Kandeel F, Kopp P, Lamonica DM, McIver B, Raeburn CD, Ridge JA, Ringel MD, Scheri RP, Shah JP, Sippel R, Smallridge RC, Sturgeon C, Wang TN, Wirth LJ, Wong RJ, Johnson-Chilla A, Hoffmann KG, Gurski LA. NCCN Guidelines Insights: Thyroid Carcinoma, Version 2.2018. J Natl Compr Canc Netw. 2018 Dec;16(12):1429-1440. doi: 10.6004/jnccn.2018.0089. PMID 30545990
- [Background] Sun C, Li Q, Hu Z, He J, Li C, Li G, Tao X, Yang A. Treatment and prognosis of anaplastic thyroid carcinoma: experience from a single institution in China. PLoS One. 2013 Nov 5;8(11):e80011. doi: 10.1371/journal.pone.0080011. eCollection 2013. PMID 24224029
- [Background] Perrier ND, Brierley JD, Tuttle RM. Differentiated and anaplastic thyroid carcinoma: Major changes in the American Joint Committee on Cancer eighth edition cancer staging manual. CA Cancer J Clin. 2018 Jan;68(1):55-63. doi: 10.3322/caac.21439. Epub 2017 Nov 1. PMID 29092098
- [Background] Subbiah V, Kreitman RJ, Wainberg ZA, Cho JY, Schellens JHM, Soria JC, Wen PY, Zielinski C, Cabanillas ME, Urbanowitz G, Mookerjee B, Wang D, Rangwala F, Keam B. Dabrafenib and Trametinib Treatment in Patients With Locally Advanced or Metastatic BRAF V600-Mutant Anaplastic Thyroid Cancer. J Clin Oncol. 2018 Jan 1;36(1):7-13. doi: 10.1200/JCO.2017.73.6785. Epub 2017 Oct 26. PMID 29072975
- [Background] Chintakuntlawar AV, Yin J, Foote RL, Kasperbauer JL, Rivera M, Asmus E, Garces NI, Janus JR, Liu M, Ma DJ, Moore EJ, Morris JC 3rd, Neben-Wittich M, Price DL, Price KA, Ryder M, Van Abel KM, Hilger C, Samb E, Bible KC. A Phase 2 Study of Pembrolizumab Combined with Chemoradiotherapy as Initial Treatment for Anaplastic Thyroid Cancer. Thyroid. 2019 Nov;29(11):1615-1622. doi: 10.1089/thy.2019.0086. PMID 31595822
- [Background] Pezzi TA, Mohamed ASR, Sheu T, Blanchard P, Sandulache VC, Lai SY, Cabanillas ME, Williams MD, Pezzi CM, Lu C, Garden AS, Morrison WH, Rosenthal DI, Fuller CD, Gunn GB. Radiation therapy dose is associated with improved survival for unresected anaplastic thyroid carcinoma: Outcomes from the National Cancer Data Base. Cancer. 2017 May 1;123(9):1653-1661. doi: 10.1002/cncr.30493. Epub 2016 Dec 27. PMID 28026871
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Chintakuntlawar AV, Rumilla KM, Smith CY, Jenkins SM, Foote RL, Kasperbauer JL, Morris JC, Ryder M, Alsidawi S, Hilger C, Bible KC. Expression of PD-1 and PD-L1 in Anaplastic Thyroid Cancer Patients Treated With Multimodal Therapy: Results From a Retrospective Study. J Clin Endocrinol Metab. 2017 Jun 1;102(6):1943-1950. doi: 10.1210/jc.2016-3756. PMID 28324060
- [Background] Lorusso L, Pieruzzi L, Biagini A, Sabini E, Valerio L, Giani C, Passannanti P, Pontillo-Contillo B, Battaglia V, Mazzeo S, Molinaro E, Elisei R. Lenvatinib and other tyrosine kinase inhibitors for the treatment of radioiodine refractory, advanced, and progressive thyroid cancer. Onco Targets Ther. 2016 Oct 20;9:6467-6477. doi: 10.2147/OTT.S84625. eCollection 2016. PMID 27799794
- [Background] Sun Y, Niu W, Du F, Du C, Li S, Wang J, Li L, Wang F, Hao Y, Li C, Chi Y. Safety, pharmacokinetics, and antitumor properties of anlotinib, an oral multi-target tyrosine kinase inhibitor, in patients with advanced refractory solid tumors. J Hematol Oncol. 2016 Oct 4;9(1):105. doi: 10.1186/s13045-016-0332-8. PMID 27716285
- [Background] Ruan X, Shi X, Dong Q, Yu Y, Hou X, Song X, Wei X, Chen L, Gao M. Antitumor effects of anlotinib in thyroid cancer. Endocr Relat Cancer. 2019 Jan 1;26(1):153-164. doi: 10.1530/ERC-17-0558. PMID 30139768
- [Background] Gunda V, Gigliotti B, Ashry T, Ndishabandi D, McCarthy M, Zhou Z, Amin S, Lee KE, Stork T, Wirth L, Freeman GJ, Alessandrini A, Parangi S. Anti-PD-1/PD-L1 therapy augments lenvatinib's efficacy by favorably altering the immune microenvironment of murine anaplastic thyroid cancer. Int J Cancer. 2019 May 1;144(9):2266-2278. doi: 10.1002/ijc.32041. Epub 2019 Jan 24. PMID 30515783
- [Background] Golden EB, Apetoh L. Radiotherapy and immunogenic cell death. Semin Radiat Oncol. 2015 Jan;25(1):11-7. doi: 10.1016/j.semradonc.2014.07.005. PMID 25481261